CLINICAL TRIAL: NCT01554306
Title: Observational Study on the Effecst of Continuous Dopaminergic Stimulation on Nocturnal Hypokinesia in Parkinson's Disease
Brief Title: Measuring the Effects of Continuous Dopaminergic Stimulation on Nocturnal Movements in Parkinson's Disease
Status: Terminated | Type: Observational
Why Stopped: difficulty to include enough subjects
Sponsor: Sleep Medicine Centre Kempenhaeghe (Other)
Responsible Party: Principal Investigator, D.A.A. Pevernagie, MD PhD, MD PhD, Sleep Medicine Centre Kempenhaeghe
Other Study IDs: 38851.091.11
Record Dates: First submitted 2012-03-05; First posted 2012-03-14 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Nocturnal Hypokinesia; Parkinsons's Disease; Rotigotine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- parkinson's disease, nocturnal hypokinesia, rotigotine

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative disorder that is characterized with motor symptoms such as hypokinesia, rigidity, tremor and postural instability. These symptoms can also be present during the night. Half of the patients with PD have difficulty turning around in bed. This nocturnal hypokinesia is considered as a possible cause of sleep problems in this population. The diagnosis nocturnal hypokinesia is based on the clinical interview. There is a need for a diagnostic devices that measures nocturnal movements, preferably in the home setting. This device can be used in the diagnostic trajectory as well in the evaluation of treatment. Recently the Dynaport Minimod (McRoberts, The Hague) has been developed to register nocturnal movements. The tri-axial accelerometer has been developed to measure position changes in the night. A validation study with actigraphy and polysomnography concluded that the Dynaport MiniMod is a valid an feasible device for assessing intensity and physical activity and changes of body position during sleep.

Nocturnal hypokinesia is treated with nocturnal dopamine. Sometimes a night-time dose of dopaminergics is adequate, but most of the time slow release dopaminergics are needed. However response fluctuations can negatively influence the treatment. In these cases continuous dopaminergic stimulation is needed, such as rotigotine. Rotigotine treats response fluctuations during the day and studies show that sleep quality measured with questionnaires improves. If the improvement of sleep quality is caused by improved bed mobility has not been studied yet. The study hypothesis is that rotigotine does not influence nocturnal hypokinesia in PD.

Objective of the study:

Primary:

• To study the effect of rotigotine on nocturnal hypokinesia

Secondary:

* To study the possibility of measuring nocturnal hypokinesia and its severity in a home setting
* To correlate improvements in sleep quality by rotigotine with changes in nocturnal hypokinesia

Study design:

We will study patients who will recieve rotigotine as a part of their usual care. During three nights, nocturnal movements are being registered with movement sensors, before treatment has started as well as after a stable medication dose of one month. We will also assess sleep quality with questionnaires.

Study population:

The study population are patients with Parkinson's disease with sleep problems caused by nocturnal hypokinesia, who will start treatment with rotigotine. Patients will be recruited in the neurology patient outdoor clinic of the Radboud University Medical Centre Nijmegen. We will ask the treating neurologist to inform us when a patient will start treatment with rotigotine. One of the researchers will contact the patient to give further information about the study. The study is a first hypothesis generating study and we will start with the inclusion of 10 patients.

Intervention (if applicable):

Primary study parameters/outcome of the study:

Position changes over the night.

Secundary study parameters/outcome of the study (if applicable):

Objective

* Degree of mobility, measured as the speed of the movements
* Total amount of movements
* Score on the motor symptom scale according to the MDS-UPDRS part III

Subjective

* Nocturnal sleep quality Excessive daytime sleepiness
* Presence of nocturnal akinesia

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic PD (defined by UK Brain Bank criteria)
* Patients who will start treatment with rotigotine
* Hoehn & Yahr stage II - IV
* Subjective sleep problems most likely caused by nocturnal hypokinesia, based on clinical interview

Exclusion Criteria:

* Other significant causes for nocturnal motor symptoms which are not dopamine-responsive
* Previous surgery for PD
* Mini- mental state examination score < 25
* Concurrent hallucination or psychosis
* History of skin hypersensitivity to adhesives or other transdermals

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Parkinson's disease with nocturnal hypokinesia based on the clinical interview who are going to start with rotigotine
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Position changes over the night. | max 1 year

SECONDARY OUTCOMES:
• Degree of mobility, measured as the speed of the movements | Max 1 year
• Total amount of movements | Max 1 year
• Score on the motor symptom scale according to the MDS-UPDRS part III | Max 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dirk AA Pevernagie, MD PhD, Study Director — Sleep Medicine Centre Kempenhaeghe
Locations (1):
- Sleep Medicine Centre Kempenhaeghe, Heeze, Netherlands